CLINICAL TRIAL: NCT03710187
Title: Hydrocortisone and Fludrocortisone Versus Hydrocortisone Alone in Critically Ill Medical Patients With Septic Shock
Brief Title: HCT+F vs. HCT Alone in Critically Ill Medical Septic Shock Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHS-CC-002
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combination (Experimental): Hydrocortisone 50 mg IV Q6h plus Fludrocortisone 50 mcg PO/PFT Q24h
  Interventions: Drug: Hydrocortisone
- Hydrocortisone only (Active Comparator): Hydrocortisone 50 mg IV Q6h
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone 50 mg IV Q6h

SUMMARY:
This study will be conducted as a single-center, prospective, open-label, randomized trial that will evaluate adult patients admitted with septic shock to the medical critical care unit (MCC). The objective of the study is to determine if the use of hydrocortisone plus fludrocortisone is associated with a faster resolution of shock (defined as 24 hours vasopressor free) when compared to the use of hydrocortisone alone in medical, critically ill septic shock patients.

DETAILED DESCRIPTION:
For three consecutive months, side 1 of the medical critical care unit (MCC1) will receive hydrocortisone alone and side 2 (MCC2) will receive the combination of hydrocortisone and fludrocortisone. After the initial three months, this will be flipped and patients admitted to MCC1 will receive the combination while patients in MCC2 will receive hydrocortisone alone for three consecutive months. This change in group assignments will occur to account for the difference in number of beds between MCC1 and MCC2, and to minimize the potential differences in patient acuity by location.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill medical patients requiring addition of stress dose steroid therapy (hydrocortisone) in addition to pressors for septic shock management during ICU stay
* Fludrocortisone administered within 24 hours after initiation of hydrocortisone if in combination therapy group

Exclusion Criteria:

* Use of fludrocortisone and/or hydrocortisone for any reason other than septic shock management during ICU stay
* Fludrocortisone/hydrocortisone initiated by any service other than critical care medicine
* Prior use of fludrocortisone/hydrocortisone at time of admission (home or outside facility)
* Patients not appropriate for study inclusion as determined by provider discretion
* Patients receiving steroid therapy not in accordance with assigned group per location (MCC1 or MCC2)
* Patients re-admitted to the MCC during the same admission and restarted on vasopressor therapy will be noted during data collection and only the initial admission will be included for analysis
* Any patient receiving greater than one dose of hydrocortisone 100 mg
* Physical or medical contraindication to receiving PO or PER FT (per feeding tube) fludrocortisone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult septic shock patients were recruited from the medical intensive care unit (MICU). Patients were recruited from November 2018 through July 2019.
Pre-assignment Details: Patients were randomized to receive HCT 50mg IV Q6h or HCT+FCT 50 mcg PO/PT daily based on admission location within the MICU. Patients were included if age 18 or older, required stress dose steroid therapy, and received fludrocortisone within 24 hours of hydrocortisone if in the combination group.
Period: Overall Study
Arm/Group | Combination | Hydrocortisone Only
Started | 41 | 43
Completed | 41 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were included in study if age 18 or older, required stress dose steroid therapy, and received fludrocortisone within 24 hours of hydrocortisone if in the combination group.
Groups:
- Combination: Hydrocortisone 50 mg IV Q6h plus Fludrocortisone 50 mcg PO/PFT Q24h
  Combination (Hydrocortisone and Fludrocortisone): Hydrocortisone 50 mg IV Q6h and Fludrocortisone 50 mg PO/PFT Q24h
- Total: Total of all reporting groups
Arm/Group | Combination | Hydrocortisone Only | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants in hydrocortisone only arm did not receive Fludrocortisone.
  Participants
    Age: <=18 years | 0 | 0 | 0
    Age: Between 18 and 65 years | 41 | 43 | 84
    Age: >=65 years | 0 | 0 | 0
    Required stress dose steroid therapy: <=18 years | 0 | 0 | 0
    Required stress dose steroid therapy: Between 18 and 65 years | 41 | 43 | 84
    Required stress dose steroid therapy: >=65 years | 0 | 0 | 0
    Fludrocortisone w/in 24 hrs of hydrocortisone: number analyzed (Participants) | 41 | 00 | 41
    Fludrocortisone w/in 24 hrs of hydrocortisone: <=18 years | 0 | 0 | 0
    Fludrocortisone w/in 24 hrs of hydrocortisone: Between 18 and 65 years | 41 | 0 | 41
    Fludrocortisone w/in 24 hrs of hydrocortisone: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 19 | 26 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 37 | 40 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Shock
Description: Hours for patient to achieve 24 hours vasopressor free
Time Frame: Up to one week
Population: Adult septic shock patients admitted to the MICU. Patients were randomized to an arm of the study based on location within the MICU.
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Combination | Hydrocortisone Only
Number analyzed (Participants) | 41 | 43
Hours | 89 [60 to 132] | 84 [56 to 125]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Combination | Hydrocortisone Only
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 0/41 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03710187/Prot_SAP_000.pdf